CLINICAL TRIAL: NCT00939718
Title: Comparison of Vitamin B12 Supplementation and SSRI to SSRI Monotherapy in Treating Depression With Low Normal B12: A Randomized Open Label trialComparison of Vitamin B12 Supplementation to SSRI Versus SSRI Antidepressant Treatment Alone
Brief Title: Comparison of Vitamin B12 Supplementation to Selective Serotonin Reuptake Inhibitor (SSRI) Versus SSRI Antidepressant Treatment Alone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Ehsan Ullah Syed ; Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 081011PSY
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Major Depressive Disorder
Keywords: depression;vitamin B12;randomized control trial
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin B12 with antidepressants (Active Comparator): Subjects in this arm will receive vitamin B12 supplement (injectable)along with their routine antidepressant treatment as prescribed by their primary physicians. subjects will be blind to their arm allocation and will receive injections in a concealed manner with injection vials covered with foil.
  Interventions: Dietary Supplement: Vitamin B12
- Placebo injections dextrose water (Placebo Comparator): Subjects in this arm will receive placebo injections which will contain only dextrose water. They will also receive 6 injections on a weekly basis and the injection vials will be covered with foil to ensure masking.
  Interventions: Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — Vitamin B12 injections containing methylcobalamin 1000 mcg given once every six months along with the routine antidepressant treatment.
  Other Names: Injection Bevidox intramuscular

SUMMARY:
While treating depression, significant numbers respond poorly to anti-depressants; one cause is vitamin B12 deficiency. The investigators are conducting an open label randomized controlled trial to investigate difference in response to SSRI monotherapy alone versus SSRI and intramuscular B12 replacement in people with low-normal B12 levels. 300 participants will be allocated to each arm of intervention at out patient clinics of the department of Psychiatry at Aga Khan University Hospital, Karachi Pakistan. Baseline and 3 month measurement of depression will be on Hamilton Rating Scale for Depression (Urdu version) and response rates compared.

DETAILED DESCRIPTION:
Vitamin B12 plays an important role in DNA synthesis and neurological function. Its deficiency is associated with hematological, neurological and psychiatric manifestations of which the latter include irritability, personality change, depression, dementia and rarely, psychosis. Recent literature has seen links between this vitamin and depression. High B12 levels in serum are associated with good treatment response, high homocysteine levels are common in folate / B12 deficiency and in those suffering from depression. Hyperhomocysteinemia may have direct effects on neurotransmitters implicated in depression.

Randomized trials have shown folate and other nutritional supplementations are strategies of atleast significant effect in treating treatment-resistant depression. Folate deficiency has also been linked with delay in treatment response as well as relapse.

To date no trial from Pakistan compares anti-depressant monotherapy with B12 augmentation in a population showing poor or partial response to first drug trial. The investigators aim to compare clinical response of SSRI-monotherapy with that of B12-augmentation in a sample of depressed patients.

Objective

To compare reduction in depression of patients with low normal B12 levels on SSRI monotherapy with patients on a combination of SSRI and Vitamin B12 supplementation.

Hypothesis There will be higher response rate among patients who will be treated with combined SSRI therapy and B12 supplementation as compared to those who will be treated with SSRI alone.

Operational Definitions Depression: Patients scoring ≥ 16 on the 17-item Hamilton Rating Scale for Depression-Urdu version (HAM-D) 24, 25 Low B12 level : (<300 pg/ml)

Design open label Trial

Setting of the Study Out patient clinics of the department of Psychiatry at Aga Khan University Hospital, Karachi Pakistan.

Duration 12 months after approval of protocol

Sample Size Calculation A total of 232 patients equally divided into two groups will achieve 90 percent power, 5 percent level of significance using one sided hypothesis and an anticipated difference in the response rate of 20 percent in the two groups with 30 percent response rate among SSRI group and atleast 50% in the combination treatment group. Considering 15 percent drop out in each group an additional sample of 36 patients equally divided into two groups will be recruited to make a total required sample of 268 patients.

Therefore sample size required for each arm would be 134.

Sampling Technique

268 consecutive patients - who fulfill the inclusion criteria given below - presenting to physicians at the PAMH Clinic will be recruited after informed consent. Consequently, 134 would be randomized to SSRI-monotherapy group and B12 augmentation group each

Method

Patients will be recruited at outpatient clinic of AKUH from among those who have received a diagnosis of major depressive disorder by a qualified psychiatrist there. After this they will be explained the research study in a simple language and will be registered after the informed consent. At this point a unique ID will be assigned to them which will be in the form of an alpha numeric code and attached to each of these ID will be a computer number which is obtained from a number series used for similar trials The research officer then will administer an Urdu version of the HAM-D scale. A blood sample of each participant will be drawn by a phlebotomist at Aga Khan University Hospital clinical laboratory. Cold chain will be maintained throughout. Those who will be fulfilling the eligibility criteria will then be recruited to the study. After recruitment these numbers will be randomized to the two arms of the study by the computer itself. The procedure will be performed by a data entry operator who will have no affiliation with the research team and will be hired on per diem basis for this purpose only. Final recruitment may take place in the next visit after the B12 levels are back. The entire process will be monitored by the research officer who will be supervised by a consultant psychiatrist at AKUH clinic who is also principal investigators. The research officer as well as the supervisor will be blind to the arm allocation and will know only codes such as Arms A and B. Participants in the monotherapy arm will only receive the SSRI. Those in B12 arm will concomitantly be administered B12 intramuscular injectable as 1000 mcg every week for 06 weeks . HAM-D scoring will be monitored at baseline and 12 weeks after the baseline.

The investigators will also be blind to the group assignment but will not be blind to the outcome assessment.The injectables will be picked up by the research officer or the patient from the main pharmacy AKUH or any designated pharmacy outlet within AKUH campus.

Any adverse effects on oral medications and injections (B12 or placebo) will be monitored and documented on a progress sheet in patient folder and treated according to the guidelines and standard of care. In case of an unfortunate rare event such as anaphylactic shock the patient will be managed according to the AKUH protocol. A crash cart will be available at the clinic all the time. The registered nurse is always present at the clinic who is ACLS certified Instruments

Hamilton Depression Rating Scale (HAM-D) 24, 25 is a 21-item, multiple-choice questionnaire that screens for severity of depression. Available in several languages, Urdu version has been translated but not clinically validated25. Therefore a pilot study will be conducted on 10% of sample size in the target population and compared with diagnosis on psychiatric interview along DSM-IV criteria for depression (gold standard).

The items comprise of cardinal and biological symptoms of depression in the first 17 items, with 3 further questions to rule out paranoia and obsessions. A score of ≥ 16 on the first 17-items correlates with clinical depression.

ELIGIBILITY:
Inclusion Criteria:

* Adults between ages 18 to 64 years who meet the criteria for a depressive episode as measured by a score of ≥ 16 on first 17 items of HAM-D (Urdu version.
* Patients with low normal B12 levels in serum (>191 but < 300 pg/ml)
* Those who will provide informed consent

Exclusion Criteria:

* Patients with concurrent unstable medical illness
* History of manic episodes or psychotic illness
* Psychotic symptoms within depressive episode

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Decline in HAM-D score of 20% or more from baseline indicating improvement in Depression. | 03 months

CONTACTS AND LOCATIONS:
Overall Officials: Anwer Siddiqui, PhD, Study Chair — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan